CLINICAL TRIAL: NCT07252674
Title: Impact of Laryngeal Mask Airway Versus Endotracheal Intubation on Mechanical Power and Postoperative Respiratory Complications in Pediatric Patients: A Prospective Observational Study
Brief Title: Comparison of Laryngeal Mask Airway and Endotracheal Intubation on Mechanical Power in Pediatric Patients
Acronym: LMA-MP
Status: Recruiting | Type: Observational
Sponsor: Konya City Hospital (Other)
Responsible Party: Principal Investigator, Esma Karaarslan, Medical Doctor (MD), Department of Anesthesiology and Reanimation, Konya City Hospital, Konya City Hospital
Other Study IDs: LMA-MP
Record Dates: First submitted 2025-11-18; First posted 2025-11-28 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-02

CONDITIONS: Mechanical Power
Keywords: Mechanical Power; Laryngeal Mask Airway; Endotracheal Intubation; Postoperative Respiratory Complications
MeSH Terms: interventions — Laryngeal Masks

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group 1: LMA Group: Group 2: ETT Group
  Interventions: Procedure: Laryngeal Mask Airway (LMA)

INTERVENTIONS:
Procedure: Laryngeal Mask Airway (LMA) — Randomization is not applied in this study. Since the research is observational in nature, the allocation of patients to the LMA or ETT groups is not performed randomly; instead, it is determined by the attending anesthesiologist based on the type of surgery, clinical requirements, and the individual characteristics of the patient. Accordingly, the choice of airway management method is not influenced by the investigators; the treatment process proceeds according to routine clinical practice, prioritizing patient safety and established clinical standards.
  Group 1: LMA Group Description: This cohort consists of pediatric patients in whom a Laryngeal Mask Airway (LMA) is used for airway management during surgery.
  Group 2: ETT Group Description: This cohort consists of pediatric patients who undergo Endotracheal Intubation (ETT) for airway management during surgery.

SUMMARY:
This prospective observational study aims to compare two commonly used airway management methods-Laryngeal Mask Airway (LMA) and Endotracheal Intubation (ETT)-in pediatric patients undergoing elective surgery under general anesthesia. The primary objective is to evaluate the impact of LMA and ETT on intraoperative mechanical power, an emerging indicator of ventilator-induced lung stress. Secondary objectives include assessing postoperative respiratory complications such as cough, hypoxemia, laryngospasm, bronchospasm, increased secretions, and breath-holding episodes. No interventions will be assigned based on a study protocol; airway management will be determined solely by clinical requirements. Routine ventilator parameters will be recorded, and mechanical power will be calculated using a validated simplified formula.

DETAILED DESCRIPTION:
This prospective, observational, single-center clinical study will be conducted in the Department of Anesthesiology and Reanimation at Konya City Hospital. The aim of the study is to compare the effects of Laryngeal Mask Airway (LMA) and Endotracheal Intubation (ETT) on intraoperative mechanical power in pediatric patients aged 2-5 years undergoing elective surgical procedures under general anesthesia. Mechanical power, calculated from routinely measured ventilator parameters, reflects the energy delivered to the respiratory system and is considered an important marker of ventilator-induced lung injury. Understanding how different airway devices influence mechanical power may contribute to improving lung-protective ventilation strategies in pediatric anesthesia.

Randomization will not be applied in this study. Airway management (LMA or ETT) will be chosen solely by the attending anesthesiologist based on clinical needs, including procedure type, expected duration, and aspiration risk. A standardized anesthesia induction and maintenance protocol will be applied to all patients. Mechanical power will be measured at two time points: (1) immediately after securing the airway and (2) at the end of surgery before emergence. Postoperative respiratory complications-including cough, hypoxemia, laryngospasm, bronchospasm, increased secretions, and breath-holding-will be systematically recorded in the Post-Anesthesia Care Unit (PACU).

To minimize observer bias, intraoperative mechanical power measurements and postoperative complication assessments will be performed by different members of the research team. No deviations from routine clinical practice will occur, and no additional interventions will be introduced. Based on the power analysis for the primary outcome, the study aims to include a total of 100 pediatric patients, with 50 patients in the LMA group and 50 patients in the ETT group.

The findings of this research are expected to provide new insights into the effects of different airway devices on mechanical power and to support the development of lung-protective anesthesia strategies in pediatric patients.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 2-5 years
* Body weight between 10-20 kg
* Patients classified as ASA physical status I-III
* Elective surgery planned under general anesthesia

Exclusion Criteria:

* Presence of severe chronic lung disease (e.g., advanced bronchopulmonary dysplasia)
* Uncontrolled or severe bronchial asthma
* Severe cardiac failure (NYHA Class III-IV)
* Diagnosis of pulmonary hypertension
* History of major lung surgery
* Severe obesity (BMI > 95th percentile)
* Children scheduled for abdominal or thoracic surgery
* Procedures expected to last longer than one hour
* Emergency surgeries
* Children and/or parents who decline participation in the study

Ages: 2 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The study population consists of pediatric patients aged 2-5 years and weighing 10-20 kg who will undergo elective surgery under general anesthesia at Konya City Hospital. Participants will be classified as ASA physical status I-III. Patients who meet all inclusion criteria and do not meet any exclusion criteria will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-11-30 (Actual); Primary Completion 2026-02-20 (Estimated); Study Completion 2026-02-25 (Estimated)

PRIMARY OUTCOMES:
Mechanical power (MP) | Mechanical power will be measured twice during surgery, as follows: MP1: Immediately after airway placement, before the start of surgery. MP2: At the end of surgery, before the initiation of emergence.
  To compare the effects of laryngeal mask airway (LMA) and endotracheal intubation (ETT) on intraoperative mechanical power (MP) in pediatric patients aged 2-5 years undergoing elective surgery under general anesthesia.
  Mechanical power (MP) will be assessed using ventilator-derived respiratory parameters (tidal volume, respiratory rate, PEEP, peak pressure, and plateau pressure). MP will be calculated using the following validated equation:
  Mechanical Power (J/min) = 0.098 × RR × VT × (PEEP + ½(Pplat - PEEP) + (Ppeak - Pplat)).

SECONDARY OUTCOMES:
Postoperative Respiratory Complications | From the start of emergence until discharge from PACU (assessed up to approximately 60 minutes).
  Respiratory complications observed during the emergence period and in the Post-Anesthesia Care Unit (PACU), including cough, breath holding, laryngospasm, bronchospasm, increased secretions, and oxygen desaturation, will be systematically recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Esma Karaarslan, MD, Principal Investigator — Konya City Hospital
Locations (1):
- Konya City Hospital, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
If data sharing is approved by the research team in the future, anonymized individual participant data (IPD) may be shared with qualified researchers upon reasonable request. Any shared data would exclude identifying information and would include only demographic variables and study-related measurements.